CLINICAL TRIAL: NCT01195129
Title: HydroCoil Cerebral Aneurysm Treatment Trial
Acronym: HCAT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to results shown by the Cerecyte Clinical Trial, HCAT stopped enrolling.
Sponsor: University of Virginia (Other)
Collaborators: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13861
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Intracerebral Aneursym
Keywords: Stent; cerebral aneursym; neurology; radiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MicroVention Hydrogel Coils (Other): FDA approved and in common use for cerebral aneurysm treatment.
  Interventions: Device: MicroVention Hydrogel coil
- Non-hydrogel coils (Active Comparator): Cerecyte or bare platinum coils (FDA approved and in common use for treatment of cerebral aneurysm).
  Interventions: Device: Non-hydrogel coils

INTERVENTIONS:
Device: MicroVention Hydrogel coil — Micro Vention Hydrogel Coils
  Arms: MicroVention Hydrogel Coils
Device: Non-hydrogel coils — Cerecyte or bare platinum coils
  Arms: Non-hydrogel coils

SUMMARY:
The study will compare clinical and angiographic outcomes in patients receiving Hydrocoil aneurysm treatment versus patients receiving non-HydroCoil aneurysm treatment.

DETAILED DESCRIPTION:
With prospective, randomized trials in progress evaluating the effectiveness of Hydrocoils and Cerecyte coils in comparison to bare platinum coils, the next step is a direct comparison of Hydrocoils and non-HydroCoils (Cerecyte or Platinum). Considering the increased costs to society of treatment with these new coils, it is essential that the benefits of the new technology are properly evaluated against the existing platinum coil technology in a scientifically valid manner.

ELIGIBILITY:
Inclusion Criteria:

1. Patient presenting with a ruptured or un-ruptured cerebral aneurysm appropriate for endovascular treatment as determined by the neurovascular team (neurosurgeon/neurointerventionalist)
2. The neurointerventionalist believes that the aneurysm can be safely treated with either Cerecyte or Hydrogel.
3. Patients between (and including) 21 and 90 years of age.
4. Patient HUNT AND HESS Grade 0-3.
5. Patient has given fully informed consent to endovascular coiling procedure. If patient cannot consent for themselves, appropriate written consent has been sought from their next of kin, or from appropriate power of attorney.
6. Aneurysm 5-20mm in maximum diameter.
7. Patient is willing and able to return for clinical evaluation and follow-up imaging evaluation (angiography or MRA) at both 6-months and 12-18 months after endovascular treatment.
8. The patient has not been previously randomized into this or another related ongoing trial.
9. The aneurysm has not previously been treated (by coiling or clipping).

Exclusion Criteria:

1. Patient has more than one aneurysm requiring treatment in the current treatment session If a patient has multiple aneurysms, but only one will be treated at the time of enrollment, they are eligible for the trial. (Additional aneurysms may be treated at a later date, and may be treated with any coil type that the operator chooses).
2. Target aneurysm has had previous coil treatment or surgically clipped.
3. Patient has an H&H score of 4 or 5 after subarachnoid hemorrhage (SAH).
4. Inability to obtain informed consent.
5. Medical or surgical co-morbidity such that the patient's life expectancy is less than 1 year.

   -

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2008-12; Primary Completion 2013-04 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Occlusion rate | 12 - 18 months
  Angiographic occlusion, improvement or no change in the post-coiling appearance of the aneurysm as judged by an independent core lab on follow-up angiography at 12-18 months after endovascular treatment.

SECONDARY OUTCOMES:
Treatment related morbidity and mortality | 12-18 months
  Treatment related morbidity and mortality, as measured by the NIH stroke scale;
Packing density | 12-18 months
  Packing density as measured by volumetric filling of the aneurysm.
Clinical outcome | 6 months
  Clinical outcome as measured by Modified Rankin Scale
Clinical Outcome | 12-18 months
  Clinical outcome as measured by the Modified Rankin scale
Re-bleed rates | 12-18 months
  Comparison of rebleed rates at 12-18 months
Re-treatment rates | 12-18 months
  Comparison of re-treatment rates at 12-18 months post treatment.
Cost of treatment | 12-18 months
  Comparison of cost of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Avery J Evans, MD, Principal Investigator — University of Virginia
Locations (11):
- United States (11):
  - Mercy Stroke Center, Carmichael, California
  - University of Southern California, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Saint Louis University, St Louis, Missouri
  - St. Luke's/Roosevelt Hospital Center, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Medical college of South Carolina, Charleston, South Carolina
  - University of Texas Southwest Medical Center, Dallas, Texas
  - The Methodist Research Institute, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia